CLINICAL TRIAL: NCT04368949
Title: Stepping-Up: Partnering with the Community to Prevent Early Mobility Decline
Acronym: Stepping-Up
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: YMCA Hamilton/Burlington/Brantford (Unknown); City of Hamilton (Unknown)
Responsible Party: Principal Investigator, Julie Richardson, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PJT-169034
Record Dates: First submitted 2020-04-23; First posted 2020-04-30 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Mobility Limitation
Keywords: Preclinical mobility limitation; Walking ability; Physical function; Task-oriented motor learning; Self-management
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stepping-Up Group (Experimental): Participants will attend one 2-hour virtual session (1-hour exercise and 1-hour SM) per week. Each class of 6-8 participants is supervised by a Physiotherapist (PT) and kinesiologist who will individually tailor the exercises for each participant.
  Interventions: Other: Stepping-Up
- TELE Group (Active Comparator): The initial telephone session will be 20-30 minutes, with subsequent weekly calls will be approximately 10 minutes.
  Interventions: Other: Telephone-Based Coaching Walking Program
- Chair-Based Yoga Group (Placebo Comparator): Participants will attend two 1-hour virtual sessions per week to ensure this group is matched for attention to STEPPING-UP.
  Interventions: Other: Chair-Based Yoga Program

INTERVENTIONS:
Other: Stepping-Up — The intervention group will receive STEPPING-UP, a virtual 12-week, multicomponent intervention that includes tailored task-oriented motor learning exercise and a mobility self-management (SM) program.
  Arms: Stepping-Up Group
Other: Telephone-Based Coaching Walking Program — The participants assigned to this group will receive a 12-week Telephone-Based Coaching Walking Program (TELE) delivered by a PT who will help participants set short and long term walking goals.
  Arms: TELE Group
Other: Chair-Based Yoga Program — Participants assigned to this group will receive a virtual 12-week Chair-Based Yoga Program (YOGA), a group-based exercise control where participants will undertake a seated exercise program that includes: warm up, seated and standing yoga poses, cool down.
  Arms: Chair-Based Yoga Group

SUMMARY:
Preclinical mobility limitations (PCML) manifest early in the process of declining mobility, and are not typically identified or acted upon by clinicians. These mobility limitations manifest as changes in how daily tasks such as walking are performed (slower speed, lower endurance). Persons in the PCML stage are at increased risk for the onset of disability and chronic disease. Persistent deterioration in mobility is a predictor of mortality and has been reported even in the absence of changes in activities of daily living over a two-year period. Further, older persons with mobility limitations, including reduced gait speed, are at risk for falls. These cumulative transitions of a person's life-long mobility form their mobility trajectory and preventing mobility decline at an early stage along this trajectory is the focus of this research initiative. This study will evaluate a novel intervention, STEPPING-UP, for improving walking ability in persons with PCML.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling
2. Age ≥55-75 years
3. PCML as assessed using a questionnaire that requires respondents to self-report difficulties with their mobility (walking 2.0km). Respondents will be considered in a stage of PCML if they report no task difficulty but report modification of task performance (i.e. modify frequency, method or time to complete the task)
4. Understanding of spoken and written English
5. Own a laptop computer, have an email address and have internet capabilities of running the video-conferencing platform, Zoom©.
6. Resident of Ontario, Canada

Exclusion Criteria:

1. A score of <11 on the MoCA 5-Minute telephone screen
2. Major illness that would prevent participation

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Walking speed | Baseline
  The 4-Metre Gait Speed Test (4MGS) is a performance-based measure of walking speed. The 4MGS test will be performed from a standing start at both a self-selected (usual) and fastest walking speed.
Change in walking speed from baseline | 12 weeks
  The 4-Metre Gait Speed Test (4MGS) is a performance-based measure of walking speed. The 4MGS test will be performed from a standing start at both a self-selected (usual) and fastest walking speed.

SECONDARY OUTCOMES:
Change in walking speed from baseline | 24 weeks
  The 4-Metre Gait Speed Test (4MGS) is a performance-based measure of walking speed. The 4MGS test will be performed from a standing start at both a self-selected (usual) and fastest walking speed.
Change in walking speed from baseline | 36 weeks
  The 4-Metre Gait Speed Test (4MGS) is a performance-based measure of walking speed. The 4MGS test will be performed from a standing start at both a self-selected (usual) and fastest walking speed.
Exercise capacity | Baseline
  2-Minute Step Test (TMST): The TMST is a test of exercise capacity that can be used as an alternative to a timed long-distance walking test when assessment space is limited. Individuals are required to march in place as quickly as possible for 2 minutes while lifting their knees to a height midway between their patella and iliac crest when standing.
Change in exercise capacity from baseline | 12 weeks
  2-Minute Step Test (TMST): The TMST is a test of exercise capacity that can be used as an alternative to a timed long-distance walking test when assessment space is limited. Individuals are required to march in place as quickly as possible for 2 minutes while lifting their knees to a height midway between their patella and iliac crest when standing.
Change in exercise capacity from baseline | 24 weeks
  2-Minute Step Test (TMST): The TMST is a test of exercise capacity that can be used as an alternative to a timed long-distance walking test when assessment space is limited. Individuals are required to march in place as quickly as possible for 2 minutes while lifting their knees to a height midway between their patella and iliac crest when standing.
Change in exercise capacity from baseline | 36 weeks
  2-Minute Step Test (TMST): The TMST is a test of exercise capacity that can be used as an alternative to a timed long-distance walking test when assessment space is limited. Individuals are required to march in place as quickly as possible for 2 minutes while lifting their knees to a height midway between their patella and iliac crest when standing.
Lower body strength | Baseline
  30-Second Chair Stand Test (CST): The 30-Second CST is used to assess lower body strength and power and is measured by the number of chair stand repetitions in a 30-second period.
Change in lower body strength from baseline | 12 weeks
  30-Second Chair Stand Test (CST): The 30-Second CST is used to assess lower body strength and power and is measured by the number of chair stand repetitions in a 30-second period.
Change in lower body strength from baseline | 24 weeks
  30-Second Chair Stand Test (CST): The 30-Second CST is used to assess lower body strength and power and is measured by the number of chair stand repetitions in a 30-second period.
Change in lower body strength from baseline | 36 weeks
  30-Second Chair Stand Test (CST): The 30-Second CST is used to assess lower body strength and power and is measured by the number of chair stand repetitions in a 30-second period.
Dual task cost | Baseline
  Difference in time between the Timed Up and Go (TUG) and the TUG Cognitive.
Change in dual task cost from baseline | 12 weeks
  Difference in time between the Timed Up and Go (TUG) and the TUG Cognitive.
Change in dual task cost from baseline | 24 weeks
  Difference in time between the Timed Up and Go (TUG) and the TUG Cognitive.
Change in dual task cost from baseline | 36 weeks
  Difference in time between the Timed Up and Go (TUG) and the TUG Cognitive.
Self-reported change in mobility | 12 weeks
  Global Mobility Change Rating: A single question, ''Since your last visit, has there been any change in your mobility?'' will be asked. The response will be made on a 11-point self-reported Likert scale: - 5 = very much worse; 0 = unchanged; 5 = very much better.
Change in self-reported change in mobility from basseline | 24 weeks
  Global Mobility Change Rating: A single question, ''Since your last visit, has there been any change in your mobility?'' will be asked. The response will be made on a 11-point self-reported Likert scale: - 5 = very much worse; 0 = unchanged; 5 = very much better.
Change in self-reported change in mobility from basseline | 36 weeks
  Global Mobility Change Rating: A single question, ''Since your last visit, has there been any change in your mobility?'' will be asked. The response will be made on a 11-point self-reported Likert scale: - 5 = very much worse; 0 = unchanged; 5 = very much better.
Balance self-efficacy | Baseline
  Activities-specific Balance Confidence (ABC) Scale: The ABC Scale is a self-report measure of balance confidence. Individuals are asked to rate their confidence in completing 16 common tasks without losing balance, on a scale from 0% (no confidence) to 100% (complete confidence).
Change in balance self-efficacy from baseline | 12 weeks
  Activities-specific Balance Confidence (ABC) Scale: The ABC Scale is a self-report measure of balance confidence. Individuals are asked to rate their confidence in completing 16 common tasks without losing balance, on a scale from 0% (no confidence) to 100% (complete confidence).
Change in balance self-efficacy from baseline | 24 weeks
  Activities-specific Balance Confidence (ABC) Scale: The ABC Scale is a self-report measure of balance confidence. Individuals are asked to rate their confidence in completing 16 common tasks without losing balance, on a scale from 0% (no confidence) to 100% (complete confidence).
Change in balance self-efficacy from baseline | 36 weeks
  Activities-specific Balance Confidence (ABC) Scale: The ABC Scale is a self-report measure of balance confidence. Individuals are asked to rate their confidence in completing 16 common tasks without losing balance, on a scale from 0% (no confidence) to 100% (complete confidence).
Mobility patterns | Baseline
  The Life-Space Assessment (LSA): The LSA measures a person's usual pattern of mobility during a 1-month period, documenting mobility based on how far and how often a person travels and any assistance required.
Change in mobility patterns from baseline | 12 weeks
  The Life-Space Assessment (LSA): The LSA measures a person's usual pattern of mobility during a 1-month period, documenting mobility based on how far and how often a person travels and any assistance required.
Change in mobility patterns from baseline | 24 weeks
  The Life-Space Assessment (LSA): The LSA measures a person's usual pattern of mobility during a 1-month period, documenting mobility based on how far and how often a person travels and any assistance required.
Change in mobility patterns from baseline | 36 weeks
  The Life-Space Assessment (LSA): The LSA measures a person's usual pattern of mobility during a 1-month period, documenting mobility based on how far and how often a person travels and any assistance required.
Knowledge, skill and confidence for self-management | 12 weeks
  Patient Activation Measure (PAM): The PAM is a 13-item measure of the patient's level of knowledge, skill and confidence for SM. An Activation Score is calculated as the sum of the 13 items. The Activation Score can then be converted into an Activation Level (Level 1 = low activation, Level 4 = high activation).
Change in knowledge, skill and confidence for self-management from baseline | Baseline
  Patient Activation Measure (PAM): The PAM is a 13-item measure of the patient's level of knowledge, skill and confidence for SM. An Activation Score is calculated as the sum of the 13 items. The Activation Score can then be converted into an Activation Level (Level 1 = low activation, Level 4 = high activation).
Change in knowledge, skill and confidence for self-management from baseline | 24 weeks
  Patient Activation Measure (PAM): The PAM is a 13-item measure of the patient's level of knowledge, skill and confidence for SM. An Activation Score is calculated as the sum of the 13 items. The Activation Score can then be converted into an Activation Level (Level 1 = low activation, Level 4 = high activation).
Change in knowledge, skill and confidence for self-management from baseline | 36 weeks
  Patient Activation Measure (PAM): The PAM is a 13-item measure of the patient's level of knowledge, skill and confidence for SM. An Activation Score is calculated as the sum of the 13 items. The Activation Score can then be converted into an Activation Level (Level 1 = low activation, Level 4 = high activation).
Balance | Baseline
  Unipedal Stance Test (UPST): The UPST is used to assess static balance. 68 Individuals are asked to stand barefoot on the limb of their choice until they (1) use their arms (i.e., uncross arms), (2) use their raised foot (i.e., move it toward or away from the standing limb or touched the floor), (3) move the weight-bearing foot to maintain their balance (i.e., rotate foot on the ground) or (4) maintain the position for a maximum of 45 seconds.
Change in balance from baseline | 12 weeks
  Unipedal Stance Test (UPST): The UPST is used to assess static balance. 68 Individuals are asked to stand barefoot on the limb of their choice until they (1) use their arms (i.e., uncross arms), (2) use their raised foot (i.e., move it toward or away from the standing limb or touched the floor), (3) move the weight-bearing foot to maintain their balance (i.e., rotate foot on the ground) or (4) maintain the position for a maximum of 45 seconds.
Change in balance from baseline | 24 weeks
  Unipedal Stance Test (UPST): The UPST is used to assess static balance. 68 Individuals are asked to stand barefoot on the limb of their choice until they (1) use their arms (i.e., uncross arms), (2) use their raised foot (i.e., move it toward or away from the standing limb or touched the floor), (3) move the weight-bearing foot to maintain their balance (i.e., rotate foot on the ground) or (4) maintain the position for a maximum of 45 seconds.
Change in balance from baseline | 36 weeks
  Unipedal Stance Test (UPST): The UPST is used to assess static balance. 68 Individuals are asked to stand barefoot on the limb of their choice until they (1) use their arms (i.e., uncross arms), (2) use their raised foot (i.e., move it toward or away from the standing limb or touched the floor), (3) move the weight-bearing foot to maintain their balance (i.e., rotate foot on the ground) or (4) maintain the position for a maximum of 45 seconds.
Health-related quality of life | Baseline
  EQ-5D-5L is a generic utility-based health related quality of life questionnaire. Respondents are asked to rate 5 dimensions of their health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The five response levels are:no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to /extreme problems (5).
Change in health-related quality of life from baseline | 12 weeks
  EQ-5D-5L is a generic utility-based health related quality of life questionnaire. Respondents are asked to rate 5 dimensions of their health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The five response levels are:no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to /extreme problems (5).
Change in health-related quality of life from baseline | 24 weeks
  EQ-5D-5L is a generic utility-based health related quality of life questionnaire. Respondents are asked to rate 5 dimensions of their health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The five response levels are:no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to /extreme problems (5).
Change in health-related quality of life from baseline | 36 weeks
  EQ-5D-5L is a generic utility-based health related quality of life questionnaire. Respondents are asked to rate 5 dimensions of their health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The five response levels are:no problems (1), slight problems (2), moderate problems (3), severe problems (4), unable to /extreme problems (5).
Self-efficacy for physical activity: | Baseline
  Participants will be asked to rate how confident they are that they could participate in moderate intensity physical activity for 150 minutes per week using a single question on a scale of 1-10. Higher values indicate greater self-efficacy.
Change in self-efficacy for physical activity from baseline | 12 weeks
  Participants will be asked to rate how confident they are that they could participate in moderate intensity physical activity for 150 minutes per week using a single question on a scale of 1-10. Higher values indicate greater self-efficacy.
Change in self-efficacy for physical activity from baseline | 24 weeks
  Participants will be asked to rate how confident they are that they could participate in moderate intensity physical activity for 150 minutes per week using a single question on a scale of 1-10. Higher values indicate greater self-efficacy.
Change in self-efficacy for physical activity from baseline | 36 weeks
  Participants will be asked to rate how confident they are that they could participate in moderate intensity physical activity for 150 minutes per week using a single question on a scale of 1-10. Higher values indicate greater self-efficacy.
Self-reported mobility | Baseline
  Mobility Assessment Tool (MAT-sf): The MAT-sf is a video-animated tool for assessing mobility. It consists of 10 animated video clips that assess an individuals' perceived level of proficiency in performing each task.
Change in self-reported mobility from baseline | 12 weeks
  Mobility Assessment Tool (MAT-sf): The MAT-sf is a video-animated tool for assessing mobility. It consists of 10 animated video clips that assess an individuals' perceived level of proficiency in performing each task.
Change in self-reported mobility from baseline | 24 weeks
  Mobility Assessment Tool (MAT-sf): The MAT-sf is a video-animated tool for assessing mobility. It consists of 10 animated video clips that assess an individuals' perceived level of proficiency in performing each task.
Change in self-reported mobility from baseline | 36 weeks
  Mobility Assessment Tool (MAT-sf): The MAT-sf is a video-animated tool for assessing mobility. It consists of 10 animated video clips that assess an individuals' perceived level of proficiency in performing each task.
Emergency room visits | Baseline to 12 weeks
  Healthcare utilization data collected using self-report self-report.
Emergency room visits | 12 weeks to 24 weeks
  Healthcare utilization data collected using self-report self-report.
Emergency room visits | 24 weeks to 36 weeks
  Healthcare utilization data collected using self-report self-report.
Hospitalizations | Baseline to 12 weeks
  Healthcare utilization data collected using self-report self-report.
Hospitalizations | 12 weeks to 24 weeks
  Healthcare utilization data collected using self-report self-report.
Hospitalizations | 24 weeks to 36 weeks
  Healthcare utilization data collected using self-report self-report.
Family doctor visits | Baseline to 12 weeks
  Healthcare utilization data collected using self-report self-report.
Family doctor visits | 12 weeks to 24 weeks
  Healthcare utilization data collected using self-report self-report.
Family doctor visits | 24 weeks to 36 weeks
  Healthcare utilization data collected using self-report self-report.
Specialist physician visits visits | Baseline to 12 weeks
  Healthcare utilization data collected using self-report self-report.
Specialist physician visits visits | 12 weeks to 24 weeks
  Healthcare utilization data collected using self-report self-report.
Specialist physician visits visits | 24 weeks to 36 weeks
  Healthcare utilization data collected using self-report self-report.
Medical tests or procedures | Baseline to 12 weeks
  Healthcare utilization data collected using self-report self-report.
Medical tests or procedures | 12 weeks to 24 weeks
  Healthcare utilization data collected using self-report self-report.
Medical tests or procedures | 24 weeks to 36 weeks
  Healthcare utilization data collected using self-report self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Richardson, PhD, Principal Investigator — McMaster University; Ayse Kuspinar, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richardson J, Kuspinar A, Sinclair S, Beauchamp M, Dufour S, Tang A, MacDermid J, Durocher E, Thabane L, Xie F, Costa A. Effect of an Online Mobility Self-Management Program on Walking Speed in Older Adults With Preclinical Mobility Limitation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 May 21;14:e72585. doi: 10.2196/72585. PMID 40397951